CLINICAL TRIAL: NCT07282379
Title: DETECTION OF ISAR-FLAGGED AT-RISK MEDICATION IN THE EMERGENCY DEPARTMENT (DISARMED)
Brief Title: Association Between Geriatric Frailty and Medication Related Problems in the Emergency Department to Help Clinical Pharmacists Prioritise Patients
Acronym: DISARMED
Status: Not yet recruiting | Type: Observational
Sponsor: Pharmacie des Hopitaux de l'Est Lemanique (Other)
Responsible Party: Sponsor
Other Study IDs: DISARMED2026
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Frailty; Emergency Department Visit; Elderly; Drug Drug Interaction; Inappropriate Drug Use
Keywords: emergency department; clinical pharmacists; elderly; frailty; ISAR; inappropriate prescription; Drug interaction; drug-related problems
MeSH Terms: conditions — Frailty; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly patients in the ED: Patients aged of 75 or more who are admitted to the emergency department
  Interventions: Other: Pharmaceutical analysis based on the Electronic Patient Record

INTERVENTIONS:
Other: Pharmaceutical analysis based on the Electronic Patient Record — After inclusion, each patient's data will be collected and analysed by the investigator in the following 5 days. The said data will be:
  * Independent variables (demographic data, laboratory results, comorbidities, home medication treatment, reason for admission)
  * The ISAR score, using the electronic patients record
  * The number of inappropriate prescriptions, using STOPP/START version 3 online tool.
  * The number of high-risk drug interactions (categories D "Consider therapy modification" and X "Avoid combination"), using Lexicomp™ Interact online tool.
  * The number of drug-related problems, using the PCNE classification version 9.1, including usual home patient's treatment as well as treatment received in the ED.
  * The likelihood of a medication-related emergency consultation, using AT-HARM 10 score.

SUMMARY:
The healthcare systems are under increasing pressure due to a rise in emergency consultations, staff shortages, an ageing population and rising costs. Emergency departments are seeing more vulnerable patients, including elderly people, who are often on multiple medications and at risk of medication errors.

To improve safety, the integration of pharmacists specialising in emergency medicine has proven beneficial: their presence in the team improves the detection of medication-related problems, speeds up and optimises treatment, reduces rehospitalisations and lowers healthcare costs. However, in most countries, these pharmacists are still rarely found in emergency departments, mainly due to a lack of resources and clinical prioritisation criteria tailored for them and adapted to this environment.

Frailty screening tools and scores, such as ISAR, can be used to identify the elderly patients most at risk, predict adverse events such as fall or mortality, and thus adapt their care in the emergency department. Indeed, elderly frail patients often take many medications and consequently are at risk of medication errors, adverse events, inappropriate prescriptions or serious drug interactions. These patients may therefore require a specialised review on their medication by clinical pharmacists when they are admitted to the emergency department, but their high number make it impossible to care for all of them.

We aim thus to evaluate the association between frailty (according to the ISAR score) and medication-related problems among elderly patients admitted to the emergency department. Researchers will examine whether this score can predict the presence of inappropriate prescribing and high-risk drug interactions. If so, pharmacists would then have a quick and easy tool to prioritise patients who would benefit most from a specialised review of their medications when they visit the emergency department.

There will not be any intervention and this study will not influence patients care. Once patients agree to participate, researchers will prospectively collect medical data from elderly patients admitted to the emergency department and analyse their medical history, home medication, reason for admission, frailty score using ISAR, and perform a pharmaceutical analysis based on these data.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 75 years admitted to the adult emergency department
* Patients able to give informed consent as documented by signature or a therapeutic representative, if applicable .

Exclusion Criteria:

* Patients initially admitted to the emergency resuscitation room.
* Patients admitted to the minor accidents and emergencies room.
* Patients admitted to the stroke unit, as they just pass through the emergency department to directly proceed to the CT-scanner.
* Missing data for proper file analysis (e.g., missing usual home medication)
* Patient's inability to sign consent and no therapeutic representative available
* Patient's refusal to sign consent
* Emergency physician's refusal to include patient for any reason.

Min Age: 75 Years | Sex: All
Age Groups: Older Adult
Study Population: The study population will consist of all geriatric patients residing in the area of the Riviera-Chablais Hospital (Rennaz, Canton of Vaud, Switzerland). This hospital cares for nearly 200,000 people and its adult emergency department receives 35,000 patients per year (20% of whom are aged 75 and over).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The rate of inappropriate prescription (PIP) as a function of their ISAR score. | At the time of their admission to the emergency department
  The rate of inappropriate prescription (PIP) will be compared as a function of their ISAR score, using Poisson regression analysis. PIPs will be defined according to the STOPP/START online tool version 3, developed for geriatric patients.
The rate of high-risk drug-drug interactions (DDIs) as a function of their ISAR score. | At the time of their admission to the emergency department
  The rate of high-risk drug-drug interactions (DDIs) will be compared as a function of their ISAR score, using Poisson regression analysis. High-risk DDIs will be detected with the Lexicomp™ Interact online tool and only categories D ("Consider therapy modification") and X ("Avoid combination") will be considered.

SECONDARY OUTCOMES:
The predictive performance of the ISAR score for the detection of PIPs and high-risk DDIs. | At the time of their admission to the emergency department.
  Determining optimal ISAR threshold for predicting medication problems further improves its use in clinical settings. If possible, sensitivity, specificity, positive predictive value, negative predictive value, and Youden index will be calculated.

OTHER OUTCOMES:
The number of drug-related problems (DRPs) in function to the ISAR score. | At the time of their admission to the emergency department.
  After pharmaceutical analysis of the electronic patient file, DRPs will be classified according to the Pharmaceutical Care Network Europe Association (PCNE) V9.
The likelihood of a medication-related emergency visit in function to the ISAR score. | At the time of their admission to the emergency department.
  The likelihood of a medication-related emergency visit will be measured with the AT-HARM 10 score. This score gives a binary result ("possibly" or "unlikely" medication-related visit) and is a useful tool to exclude patients who are unlikely to be admitted due to a medication issue.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Riviera-Chablais (Vaud-Valais), service des urgences, Rennaz, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
If patients give their consent for data re-utilisation (consent signature independent from their inclusion in the study), demographic data and all individual outcomes (ISAR score, inappropriate prescriptions, high-risk drug interactions, drug-related problems, AT-HARM10 score) will be shared. All data will be anonymised and shared in a secure format (CSV).
Supporting Information: Study Protocol
Time Frame: IPD data will be available 6 months after publication of the first study results and for 10 years
Access Criteria: Data will be accessible to external researchers, regulatory bodies, and authorized entities under the following conditions:
  Formal request submission detailing the project and data usage. Access granted if the request meets ethical, scientific, and confidentiality criteria.
URL: https://olos.swiss/portal/home

REFERENCES:
- [Result] Zautra A, Hempel A. Subjective well-being and physical health: a narrative literature review with suggestions for future research. Int J Aging Hum Dev. 1984;19(2):91-110. doi: 10.2190/a9rb-7d02-g77k-m3n6. PMID 6394508
- [Result] Mowri HO, Patsch JR, Gotto AM Jr, Patsch W. Apolipoprotein A-II influences the substrate properties of human HDL2 and HDL3 for hepatic lipase. Arterioscler Thromb Vasc Biol. 1996 Jun;16(6):755-62. doi: 10.1161/01.atv.16.6.755. PMID 8640403
- [Result] McCusker J, Bellavance F, Cardin S, Trepanier S, Verdon J, Ardman O. Detection of older people at increased risk of adverse health outcomes after an emergency visit: the ISAR screening tool. J Am Geriatr Soc. 1999 Oct;47(10):1229-37. doi: 10.1111/j.1532-5415.1999.tb05204.x. PMID 10522957
- [Result] Ellis B, Carpenter CR, Lowthian JA, Mooijaart SP, Nickel CH, Melady D. Statement on Minimum Standards for the Care of Older People in Emergency Departments by the Geriatric Emergency Medicine Special Interest Group of the International Federation for Emergency Medicine. CJEM. 2018 May;20(3):368-369. doi: 10.1017/cem.2017.426. Epub 2018 Jan 23. No abstract available. PMID 29357950
- [Result] Almarsdottir AB, Haq R, Norgaard JDSV. Prioritizing patients for medication review by emergency department pharmacists: a multi-method study. Int J Clin Pharm. 2023 Apr;45(2):387-396. doi: 10.1007/s11096-022-01515-3. Epub 2022 Dec 5. PMID 36469215
- [Result] Bamps J, Lelubre S, Cauchies AS, Devillez A, Almpanis C, Patris S. Identification of seniors at risk (ISAR) score and potentially inappropriate prescribing: a retrospective cohort study. Int J Clin Pharm. 2024 Dec;46(6):1345-1351. doi: 10.1007/s11096-024-01766-2. Epub 2024 Jul 2. PMID 38954078
- See also: Web page of the hospital pharmacy conducting the study (PHEL) and describing all current research projects summaries. — https://www.phel.ch/jcms/phel_10754/projets